CLINICAL TRIAL: NCT01394133
Title: Impact of Menstrual Cycle on Antiretroviral Pharmacokinetics in HIV-Infected Women
Status: Withdrawn | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Jennifer King, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: F10102815; 1K23AI074390-01A2 (NIH)
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infected
Keywords: HIV Infected Women
MeSH Terms: interventions — Tenofovir; Emtricitabine; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5 mL of plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV+ Female: HIV infected women between 21-40 years of age, not receiving oral contraceptives.
  Interventions: Drug: Tenofovir, Emtricitabine, Atazanavir, Ritonavir

INTERVENTIONS:
Drug: Tenofovir, Emtricitabine, Atazanavir, Ritonavir — Women will be receiving Tenofovir 300mg, Emtricitabine 200mg, Atazanavir 300mg, Ritonavir 100mg, one dose on 2 separate visits. These medications will not be prescribed from the physician and not provided by the study.

SUMMARY:
Data suggests that women taking drugs to treat human immunodeficiency virus (HIV) have higher amounts of drugs in their body compared with men taking the same dose of anti-HIV drugs. The reason for this higher drug exposure has not yet been determined. The primary purpose of this study is to examine whether a pharmacokinetics (factors that determine the amount of drug in the body) of anti-HIV drugs change during different phases of the menstrual cycle in women and ultimately result in higher amounts of drug in the body compared with men. In other words, we plan to examine whether changes in sex hormones throughout the menstrual cycle affect the amount of anti-HIV drugs in HIV infected women. The antiretroviral drugs atazanavir, ritonavir, tenofovir and emtricitabine will be studied.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive females between 21-40 years of age.
* Subjects must be receiving anti-HIV regimen consisting of tenofovir, emtricitabine, atazanavir, and ritonavir for a minimum of 4 weeks prior to the study.
* Subjects must have regular menstrual cycle (period), define at least 10 cycles a year, occurring approximately every 28 days+/- 4 days and cycle length varying by not more than 7 days.

Exclusion Criteria:

* Subjects can not be breast feeding, pregnant, or taking oral contraceptives (birth control pills) for at least 3 months prior to the study.
* Subjects may not have the intrauterine device (IUD), Mirena, in place to prevent pregnancy.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-infected women will be selected from the primary care office
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
PK parameters | 28 days
  The area under the concentration time curve and minimum concentration for tenofovir, emtricitabine, atazanavir and ritonavir

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States